CLINICAL TRIAL: NCT01204021
Title: Managing Stress and Social Ties for Health Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AG028748-01-SST
Record Dates: First submitted 2010-01-25; First posted 2010-09-17 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Stress
Keywords: Stress; loneliness; social isolation; autonomic activity; inflammation; Perceived social isolation; Chronic stress
MeSH Terms: conditions — Social Isolation; Inflammation | interventions — Tai Ji; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi Chih (Experimental): 12 weeks of physical exercise in the form of Tai Chi Chih
  Interventions: Behavioral: Tai Chi Chih
- Stress Education Control (Active Comparator): Stress management education
  Interventions: Behavioral: Stress Education Control

INTERVENTIONS:
Behavioral: Tai Chi Chih — 12 weeks of weekly classes of Tai Chi Chih
  Other Names: Tai Chi; exercise; relaxation
  Arms: Tai Chi Chih
Behavioral: Stress Education Control — Weekly meetings, for 2 hours for 12 weeks discussing issues related to stress education.
  Other Names: stress education; stress information
  Arms: Stress Education Control

SUMMARY:
There has been a dramatic rise from 46% to 59% in the percentage of households with only 1-2 people from 1970 to 2000. A 40% increase in the number of people living alone is projected for 2010. Social isolation is consistently one of the strongest predictors mortality in older adults. Recent research is demonstrating that stress plays an important role linking social isolation with poor health. Socially isolated older adults are more likely to feel chronically stressed and overwhelmed with everyday life demands. Furthermore, isolated adults respond to stress differently, both psychologically and physiologically. Socially isolated and lonely older adults show long-term elevations in "inflammatory cytokines", which are signaling molecules related by immune cells. These Inflammatory cytokines play a role in a number of age-related diseases including cardiovascular disease, type-2 diabetes and arthritis. Novel, readily useable interventions aimed at decreasing isolation and "re-calibrating" stress responses might be helpful to older adults.

Tai Chi is an ancient Chinese form of calisthenics that promotes relaxation and decreases feelings of stress and as such, it may be a useful intervention for socially isolated, stressed older adults. However, its effects on stress responses are unknown. Tai Chi Chih (TCC) is a simplified, manualized, readily exportable form of Tai Chi particularly well-suited for older adults. This proposed study will test the effects of a TCC intervention with socially isolated older adults on loneliness, stress and health outcomes, including inflammatory assessment. Tai Chi-naïve participants who perceive themselves as socially isolated, as measured by the UCLA Loneliness Scale will be randomized to receive either Tai Chi or education control for a 12-week period. Subjects will undergo pre- and post-intervention stress assessment, including exposure to a psychological stress task, to assess whether Tai Chi affects how subjects physiologically and psychologically respond to stress.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 60 years old
* Have not done Tai Chi before
* Live in Los Angeles area
* Socially isolated
* Women must be post menopausal

Exclusion Criteria:

* Any physical debility that limits Tai Chi performance;
* Cognitive impairment (< 23 on the Mini-Mental State Exam);
* Current or recent history of smoking
* Immune suppression resulting from neoplastic disease
* Corticosteroid use or other therapy
* Significant underlying illness that would interfere or prevent completion of the study
* Acute conditions (e.g. viral infection w/in 2 weeks) that might confound interpretation of inflammatory data
* Current or recent (within 1 month) use of illicit drugs.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | 4-8 months

SECONDARY OUTCOMES:
Autonomic Activity and inflammatory signalling | 4-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarosh J Motivala, Ph.D., Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Result] Black DS, Irwin MR, Olmstead R, Ji E, Crabb Breen E, Motivala SJ. Tai chi meditation effects on nuclear factor-kappaB signaling in lonely older adults: a randomized controlled trial. Psychother Psychosom. 2014;83(5):315-7. doi: 10.1159/000359956. Epub 2014 Aug 6. No abstract available. PMID 25116908